CLINICAL TRIAL: NCT06810882
Title: Intravenous Versus Perineural Ondansetron as an Adjuvant in Autonomic Neural Blockade for Laparoscopic Sleeve Gastrectomy: A Two-Center, Randomized, Double-Blind, Non-inferiority Trial
Brief Title: Intravenous Versus Perineural Ondansetron for Laparoscopic Sleeve Gastrectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, lecturer of anesthesiology, surgical intensive care and pain medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR1032/1/25
Record Dates: First submitted 2025-01-27; First posted 2025-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ondansetron; Laparoscopic; Gastrectomy
Keywords: Ondansetron; Laparoscopic; Gastrectomy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Perineural ondansetron group (Experimental): Para-gastric autonomic neural blockade will be performed (after separation of the stomach and performing the methylene blue leak test) using 20 ml solution containing 18 ml bupivacaine 0.5% plus 2 ml (4 mg) ondansetron. At the same time, 15 ml saline will be injected slowly IV over 15 minutes.
  Interventions: Drug: Perineural ondansetron
- Intravenous ondansetron group (Active Comparator): Para-gastric autonomic neural blockade will be performed (after separation of the stomach and performing the methylene blue leak test) using 20 ml solution containing 18 ml bupivacaine 0.5% plus 2 ml saline. At the same time, 4 mg (2 ml) ondansetron mixed with 13 ml saline (total 15 ml) will be slowly injected IV over 15 minutes.
  Interventions: Drug: Intravenous ondansetron

INTERVENTIONS:
Drug: Perineural ondansetron — Para-gastric autonomic neural blockade will be performed (after separation of the stomach and performing the methylene blue leak test) using 20 ml solution containing 18 ml bupivacaine 0.5% plus 2 ml (4 mg) ondansetron. At the same time, 15 ml saline will be injected slowly IV over 15 minutes.
  Arms: Perineural ondansetron group
Drug: Intravenous ondansetron — Para-gastric autonomic neural blockade will be performed (after separation of the stomach and performing the methylene blue leak test) using 20 ml solution containing 18 ml bupivacaine 0.5% plus 2 ml saline. At the same time, 4 mg (2 ml) ondansetron mixed with 13 ml saline (total 15 ml) will be slowly injected IV over 15 minutes.
  Arms: Intravenous ondansetron group

SUMMARY:
This prospective randomized non-inferiority study will be conducted to compare the analgesic anti-emetic effects of intravenous ondansetron versus perineural ondansetron in patients undergoing laparoscopic sleeve gastrectomy.

DETAILED DESCRIPTION:
Obesity and its associated disorders have significant implications for health, resulting in heightened productivity loss and reduced life expectancy while also negatively impacting the quality of life of patients. Surgical intervention is the most effective way to achieve sustainable weight loss in patients with obesity and to alleviate the associated comorbidities. Despite the current availability of minimally invasive bariatric surgical treatments, postoperative pain remains a significant issue. Vagal and sympathetic afferent signals originating from the gastrointestinal system stimulate the vomiting center, causing nausea and vomiting. Paragastric autonomic neural blockade (PANB) is a new method performed by injecting local anesthetic material into three to four separate points along the border between the lesser omentum and the stomach (from the esophagogastric junction to the distal antrum), the hepatoduodenal ligament, and the area covering the left gastric artery. This procedure aims to prevent visceral pain and symptoms of nausea and vomiting. Ondansetron is a serotonin receptor (5-HT3) antagonist used commonly to manage postoperative nausea and vomiting (PONV) through intravenous (IV) injection. It also has a local anesthetic effect and many studies used it as adjuvant in various regional anesthetic techniques. In this study, investigators will compare the combined antiemetic analgesic effects of IV and perineural (adjuvant to the local anesthetic bupivacaine in PANB) ondansetron. The investigators hypothesized that perineural administration of ondansetron will be non-inferior to the IV route regarding prophylaxis against PONV, and will provide superior postoperative analgesic effects by its local anesthetic enhancing action.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex
* American Society Anesthesiologists physical (ASA) status II-III
* age between 18-65 years old
* Body mass index (BMI) >35 kg/m2 with comorbidity or > 40 kg/m2 -- undergoing laparoscopic sleeve gastrectomy with intraoperative surgeon performed laparoscopic paragastric autonomic neural blockade..

Exclusion Criteria:

* Allergy to experimental drugs.
* Known to have long QT, previous history of postoperative nausea and vomiting
* Abuse of alcohol, analgesia, or sedative antidepressant drugs
* Chronic pain disorders
* History of previous upper gastrointestinal system surgery, those with surgery-related complications during or after surgery.
* Liver or kidney failure
* Performance of concomitant procedures in addition to laparoscopic sleeve gastrectomy
* Anesthetic complications that may alter the postoperative management protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2025-02-16 (Actual); Primary Completion 2026-12-16 (Estimated); Study Completion 2026-12-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of vomiting in the early 8 hours after surgery. | 8 hours after surgery.
  Any attack of vomiting will be recorded for all patients.
Degree of postoperative pain at 1 hour after surgery as measured by the numerical rating scale pain score. | 1 hour after surgery.
  Numerical rating scale pain score (NRS) ranges from 0 = no pain to 10= worst pain.

SECONDARY OUTCOMES:
Incidence of postoperative nausea and vomiting at 1 h, 8 h, and at 24 hours after surgery. | 24 hours after surgery.
  Any attack of nausea and vomiting will be recorded for all patients. Numerical rating scale from 0 (no nausea) to 10 (worst nausea) will be used to assess the severity of nausea.
Number of rescue anti-emetic doses in the first postoperative day. | 24 hours after surgery.
  Routine anti-emetics will be given every 8 hours in the form of IV metoclopramide 10 mg. Rescue anti-emetic medication in the form of ondansetron 8 mg slowly IV will be given. The total required dose and number of ondansetron boluses will be recorded.
Postoperative pain scores at 4 h, 8 h, and 24 hour after surgery. | 24 hours after surgery.
  Numerical rating scale pain score (NRS) ranges from 0 = no pain to 10= worst pain will be used to evaluate pain scores after surgery.
Time to first rescue opioid analgesic. | 24 hours after surgery.
  opioid dose will be given to patients with pain score ≥ 4.
Total opioid dose in the first day after surgery. | 24 hours after surgery.
  opioid dose will be given to patients with pain score ≥ 4.
Patient satisfaction | 24 hours after surgery.
  Likert-type scale of 0-5 points will assess satisfaction before discharge from the hospital .

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University Hospitals, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: After completion of the study.
Access Criteria: The data will be available upon reasonable request from the corresponding author.